CLINICAL TRIAL: NCT06288958
Title: Quality of Life in Children With Cerebral Palsy: the Impact of Social Participation, Motor and Cognitive Levels
Brief Title: Quality of Life in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Principal Investigator, Giuseppina Sgandurra, MD, PhD, IRCCS Fondazione Stella Maris
Other Study IDs: Fondazione Stella Maris
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Unilateral and Bilateral Cerebral Palsy
Keywords: Cerebral Palsy; Quality of Life; Social participation; Cognitive Functioning; Motor Skills; Background Factors
MeSH Terms: conditions — Cerebral Palsy | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Cerebral Palsy: Children aged 4 to 12 with CP diagnosis
  Interventions: Other: Quality of Life and social participation in Italian children with CP

INTERVENTIONS:
Other: Quality of Life and social participation in Italian children with CP — CP-QOL and PEM-CY questionnaires are fulfilled by families of children.

SUMMARY:
Cerebral Palsy (CP) is an umbrella term that defines a group of permanent disorders of movement and posture, happening during the developing foetal or infant brain. In addition to the main motor symptoms, other clinical disturbances are associated. CP represents a clinical condition with an impact in Quality Of Life (QOL) and social participation, as reported in different countries. QOL is a multidimensional construct defined as "an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards, and concerns" (WHOQOL, 1998).

In order to best capture the peculiarities of CP, specific questionnaires were carried out to analyse the QOL in this clinical population. The Cerebral Palsy Quality of Life Questionnaire for Children (CP QOL-Child) is an internationally recognized CP-specific instrument based on the International Classification of Functioning, Disability and Health (ICF) framework. Many studies have used this instrument, showing a lower QOL in children with CP compared to their typical developing peers. In literature, several studies have shown that children with CP are at risk of experiencing activity limitations and participation restriction and which can potentially affect their QOL. Participation in daily-life activities, defined as a person's "involvement in a life situation," and participation restriction, characterised as "problems an individual may experience in involvement in life situations" (ICF, World Health Organization, 2001). Studies aimed at describing participation in daily-life activities in CP have consistently found lower frequencies and fewer activities in children and adolescents with CP. In order to gain an overall picture of the QOL and participation of children and adolescents with CP, several studies underline the importance of analysing other background factors, such as motor and cognitive functioning, pain perception, and individual characteristics.

The present study aims to deeper understand the perception of QOL and social participation in a group of Italian children with CP, as reported by their parents, using two commonly used questionnaires in the CP population (CP-QOL and PEM-CY). In addition, this study aims to explore the roles of specific clinical variables, such as motor function and cognitive level, on parental perceptions of QOL, in the development of QOL and participation.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is defined as "a group of permanent disorders of movement and posture occurring in the developing foetal or infant brain" (Rosenbaum et al., 2007). Various clinical disturbances, including behavior, cognition, communication, sensation perception, epilepsy, musculoskeletal problems, are also associated. CP represents a clinical condition with an impact in Quality Of Life (QOL) and social participation, as reported in different countries (Böling et al., 2016; Omura et al., 2018). Quality of life (QOL) is a multidimensional construct defined as "an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards, and concerns" (WHOQOL, 1998). QOL concerns several domains such as material conditions, health status, functional abilities, social interactions, and emotional well-being. In the case of children and adolescents, these aspects can be assessed by gathering information from the children themselves or their parents. The literature frequently documents notable differences between the quality of life (QOL) reports of children and their parents. In many instances, children and adolescents tend to express higher QOL assessments across different domains when compared to the evaluations provided by their caregivers (Davis et al., 2009). Parental distress also plays a crucial role in influencing their perception of their child's condition.

Given the particularity of CP and the variety of associated disorders, specific questionnaires were developed to analyse the QOL in this clinical population, in order to deeper understand the difficulties that arise. An example is the Cerebral Palsy Quality of Life Questionnaire for Children (CP QOL-Child), it is an internationally recognized CP-specific instrument based on the International Classification of Functioning, Disability and Health (ICF) framework. It was developed by an international, multidisciplinary team of clinical and child health researchers in collaboration with parents and children with CP and has been used in various countries. Many studies, using this instrument, have observed that children with CP show a good level of QOL, but lower than typically population (Radsel et al., 2016).

Furthermore, it has been shown in the literature that children with CP often experience restriction in participation and activities compared to their peers, these limitations may contribute to affecting QOL of this clinical population. Participation in daily-life activities, defined as a person's "involvement in a life situation," and participation restriction, characterised as "problems an individual may experience in involvement in life situations" (ICF, World Health Organization, 2001). Several studies, exploring daily functioning in social and home activities and the relationship between the individual and their environment, found lower participation in children and adolescents with CP respect to their peers. The level of participation seems to be a factor that influences the QOL of this clinical population. In order to better comprehend QOL and social participation in children and adolescents with CP, it is important analyse different background factors, such as motor functioning, pain perception, and individual characteristics (Makris et al., 2021) There is widespread consensus in the literature on the potential predictive role of cognitive functioning in QOL and social participation, although there are few studies on the impact of intellectual disability on the QOL of children and adolescents with CP. The present study aims to deeper understand the perception of QOL and social participation of a group of Italian children with CP. To pursue this, their parents complete the CP QOL-Child Primary Caregiver and PEM-CY questionnaires, commonly used in the CP population. In addition, this study aims to explore the roles of specific clinical variables, such as motor function and cognitive level, on parental perceptions of QOL, in the development of QOL and participation. For this reason, psychological assessment is conducted to evaluate intellectual abilities and motor assessment to describe the manual ability and gross motor skills and the independence in daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Children with confirmed diagnosis of CP

Exclusion Criteria:

* None

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Cerebral Palsy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Score of CP-QOL Child questionnaire | Months 1-32
  The CP QOL-Child questionnaire (caregiver-proxy version) assesses the QOL of children aged 4 to 12 years (Waters et al., 2006, Davis et al., 2009). This questionnaire comprises 66 items and evaluates seven domains of QOL, including Social Wellbeing and Acceptance, Functioning, Participation and Physical Health, Emotional Wellbeing and Self-esteem, Access to Services, Pain and the Impact of Disability, and Family Health. Most of the items start with the question: "How do you think your child feels about...?" using a nine-point rating scale ranging from 1 (very unhappy) to 9 (very happy). Item ratings were transformed to a 0-100 scale, with the mean of item values computed for each domain.

SECONDARY OUTCOMES:
Score of PEM-CY questionnaire | Months 1-32
  The Participation and Environment Measure for Children and Youth (PEM-CY; Coster, Law, & Bedell, 2010) is a reliable and valid instrument for parent/caregiver reporting, designed to assess children's participation and their environment in three distinct settings: home, school, and the community. In the first section of the questionnaire parents asked to indicate how frequently their child has participated in specific activities in the last four months, how much he was involved and their change desire in child's participation. The last section investigates the impact of certain environmental features and the availability of resources. Response options are based on an 8- or 5-point scale or on a yes or no choice, scores are expressed as an average or percentage.
Scores of Wechsler Intelligence scales | Months 1-32
  Verbal and Non verbal intelligence indices are obtained by the Italian version of Wechsler Intelligence Scale for Children - Fourth Edition (VCI and PRI, WISC-IV, Wechsler, 2003) for 6- to 16-year-old children; the Italian version of Wechsler Preschool and Primary Scale for Intelligence - Third edition (VIQ and PIQ, WPPSI-III, Wechsler, 2002) or - Fourth Edition (VCI and PRI, WPPSI-IV, Wechsler, 2012) for 3- to 7-year-old children were administered.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppina Sgandurra, MD, PhD, Principal Investigator — IRCCS Fondazione Stella Maris
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Boling S, Varho T, Kiviranta T, Haataja L. Quality of life of Finnish children with cerebral palsy. Disabil Rehabil. 2016;38(7):683-8. doi: 10.3109/09638288.2015.1061607. Epub 2015 Jun 29. PMID 26119576
- [Background] Omura J, Fuentes M, Bjornson K. Participation in Daily Life: Influence on Quality of Life in Ambulatory Children with Cerebral Palsy. PM R. 2018 Nov;10(11):1185-1191. doi: 10.1016/j.pmrj.2018.05.010. Epub 2018 May 18. PMID 29783065
- [Background] Bugusan S, Kahraman A, Elbasan B, Mutlu A. Do adolescents with cerebral palsy agree with their caregivers on their participation and quality of life? Disabil Health J. 2018 Apr;11(2):287-292. doi: 10.1016/j.dhjo.2017.10.009. Epub 2017 Oct 24. PMID 29100958
- [Background] Davis E, Mackinnon A, Waters E. Parent proxy-reported quality of life for children with cerebral palsy: is it related to parental psychosocial distress? Child Care Health Dev. 2012 Jul;38(4):553-60. doi: 10.1111/j.1365-2214.2011.01267.x. Epub 2011 Jun 15. PMID 21671983
- [Background] Shelly A, Davis E, Waters E, Mackinnon A, Reddihough D, Boyd R, Reid S, Graham HK. The relationship between quality of life and functioning for children with cerebral palsy. Dev Med Child Neurol. 2008 Mar;50(3):199-203. doi: 10.1111/j.1469-8749.2008.02031.x. Epub 2008 Jan 21. PMID 18215191
- [Background] Radsel A, Osredkar D, Neubauer D. Health-related quality of life in children and adolescents with cerebral palsy. Zdr Varst. 2016 Jul 28;56(1):1-10. doi: 10.1515/sjph-2017-0001. eCollection 2017 Mar 1. PMID 28289457
- [Background] Majnemer A, Shevell M, Law M, Birnbaum R, Chilingaryan G, Rosenbaum P, Poulin C. Participation and enjoyment of leisure activities in school-aged children with cerebral palsy. Dev Med Child Neurol. 2008 Oct;50(10):751-8. doi: 10.1111/j.1469-8749.2008.03068.x. PMID 18834388
- [Background] Mc Manus V, Corcoran P, Perry IJ. Participation in everyday activities and quality of life in pre-teenage children living with cerebral palsy in South West Ireland. BMC Pediatr. 2008 Oct 31;8:50. doi: 10.1186/1471-2431-8-50. PMID 18976459
- [Background] Milicevic M, Nedovic G. Comparative study of home and community participation among children with and without cerebral palsy. Res Dev Disabil. 2018 Sep;80:74-83. doi: 10.1016/j.ridd.2018.06.010. Epub 2018 Jun 27. PMID 29957491
- [Background] Michelsen SI, Flachs EM, Damsgaard MT, Parkes J, Parkinson K, Rapp M, Arnaud C, Nystrand M, Colver A, Fauconnier J, Dickinson HO, Marcelli M, Uldall P. European study of frequency of participation of adolescents with and without cerebral palsy. Eur J Paediatr Neurol. 2014 May;18(3):282-94. doi: 10.1016/j.ejpn.2013.12.003. Epub 2013 Dec 25. PMID 24412031
- [Background] Imms C, Reilly S, Carlin J, Dodd K. Diversity of participation in children with cerebral palsy. Dev Med Child Neurol. 2008 May;50(5):363-9. doi: 10.1111/j.1469-8749.2008.02051.x. Epub 2008 Mar 18. PMID 18355337
- [Background] Engel-Yeger B, Jarus T, Anaby D, Law M. Differences in patterns of participation between youths with cerebral palsy and typically developing peers. Am J Occup Ther. 2009 Jan-Feb;63(1):96-104. doi: 10.5014/ajot.63.1.96. PMID 19192732
- [Background] Majnemer A, Shikako-Thomas K, Schmitz N, Shevell M, Lach L. Stability of leisure participation from school-age to adolescence in individuals with cerebral palsy. Res Dev Disabil. 2015 Dec;47:73-9. doi: 10.1016/j.ridd.2015.08.009. Epub 2015 Sep 2. PMID 26342327
- [Background] Almasri NA, Alquaqzeh FA. Determinants of Quality of Life of Children and Adolescents with Cerebral Palsy: A Systematic Review. Phys Occup Ther Pediatr. 2023;43(4):367-388. doi: 10.1080/01942638.2022.2162358. Epub 2023 Jan 1. PMID 36588347
- [Background] Pagliano E, Casalino T, Mazzanti S, Bianchi E, Fazzi E, Picciolini O, Frigerio A, Rossi A, Gallino F, Villani A, Landi N, Roberti L, Militerni R, Di Brina C, Tornetta L, Martielli M, Brizio M, Rodocanachi M, Tessarollo V, Galli J, Dusi E, Meschini L, Malinconico E, Baranello G, Anderloni A, Fedrizzi E. Being adults with cerebral palsy: results of a multicenter Italian study on quality of life and participation. Neurol Sci. 2021 Nov;42(11):4543-4550. doi: 10.1007/s10072-021-05063-y. Epub 2021 Feb 23. PMID 33624178
- [Background] Blasco M, Garcia-Galant M, Laporta-Hoyos O, Ballester-Plane J, Jorba-Bertran A, Caldu X, Miralbell J, Alonso X, Melendez-Plumed M, Toro-Tamargo E, Gimeno F, Pueyo R. Factors Related to Quality of Life in Children With Cerebral Palsy. Pediatr Neurol. 2023 Apr;141:101-108. doi: 10.1016/j.pediatrneurol.2023.01.006. Epub 2023 Jan 18. PMID 36805966
- [Background] Makris T, Dorstyn D, Crettenden A. Quality of life in children and adolescents with cerebral palsy: a systematic review with meta-analysis. Disabil Rehabil. 2021 Feb;43(3):299-308. doi: 10.1080/09638288.2019.1623852. Epub 2019 Jun 10. PMID 31180733